CLINICAL TRIAL: NCT01464918
Title: Safety and Efficacy of Using MASTER, a Novel Robotics Enhanced Endosurgical System to Perform Endoscopic Submucosal Dissection in Human
Brief Title: Safety and Efficacy of Using MASTER to Perform Endoscopic Submucosal Dissection in Human
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Apollo Gleneagles Hospitals, Kolkata (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E11/058
Record Dates: First submitted 2011-10-30; First posted 2011-11-04 (Estimated); Last update posted 2011-11-04 (Estimated); Status verified 2011-10

CONDITIONS: Gastric Cancer; Colon Cancer
Keywords: gastric cancer; colon cancer; endoscopic submucosal dissection
MeSH Terms: conditions — Stomach Neoplasms; Colonic Neoplasms | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ESD using the MASTER device (Experimental): Endoscopic submucosal dissection of gastric/colon cancer using the device, MASTER
  Interventions: Device: Endoscopic submucosal dissection (ESD) using device, MASTER

INTERVENTIONS:
Device: Endoscopic submucosal dissection (ESD) using device, MASTER — Performing endoscopic submucosal dissection (ESD)of the gastric/colon cancer using the device, MASTER

SUMMARY:
This trial is to evaluate the safety and efficacy of using MASTER, a robotics enhanced endosurgical system to perform endoscopic submucosal dissection (ESD) of gastric/colon cancer in human.

DETAILED DESCRIPTION:
This trial is to evaluate the safety and efficacy of using MASTER, a novel robotics enhanced endosurgical system to perform endoscopic submucosal dissection (ESD) of gastric/colon cancer in human. The MASTER is a master-and-slave robotic system that is deployed through a standard dual-channel therapeutic endoscope. It introduces robotic control of endoscopic surgical tools and tasks through an ergonomic human-machine interface built around the original endoscopic paradigm. In doing so, it separates control of instrumental motion from that of endoscopic movement such that surgical tasks may be independently executed by a second operator via a human-machine interface. With it, endoscopically deployed instruments can be independently controlled, allowing thus bimanual coordination of effector instruments to facilitate actions such as retraction/exposure, traction/countertraction, approximation and dissection of tissue. Using the MASTER, operational dexterity is increased, thus making it easier for the operator to perform the ESD procedure as compared with using the conventional endoscope. This study will measure the ease of using the MASTER to perform the various surgical tasks involved in the ESD procedure, the time taken to perform the procedure, and record complications, if any, occurred during and after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* patient diagnosed with early gastric or colon cancer, is deemed suitable to undergo endoscopic submucosal dissection and is able/willing to give informed consent.

Exclusion Criteria:

* case is deemed not suitable for endoscopic submucosal dissection
* is on warfarin or other blood thinning agents and those with bleeding disorders
* has uncorrected coagulopathy or severe thrombocytopenia precluding biopsy
* has serious co-morbidities such as heart disease, renal impairment and cancer
* has recently underwent surgery or has a personal history of stomach/colon cancer or surgery
* is unable/unwilling to give informed consent
* is pregnant or breast-feeding women patients who cannot undergo gastroscopies

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Total time taken to complete the ESD procedure | Participants will be followed for the duration of the operation, an expected average of 3 hours
  The total time spent from docking of MASTER to end of submucosal dissection

SECONDARY OUTCOMES:
Measure of ease of performing the ESD procedure | Participants will be followed for the duration of the operation, an expected average of 3 hours
  Measure ease of grasping, retraction, and triangulation of robotics end-effectors during the ESD procedure. Measures are rated as "excellent, good, or poor".
Safety | From start of operation of the ESD procedure, assessed up to 7 days after the procedure
  Any procedure-related complications that occurs from start ofthe ESD procedure up to 7 days after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Khek Yu Ho, MBBS; MD, Principal Investigator — National University Hospital, Singapore
Locations (3):
- Prince of Wales Hospital, Shatin, Hong Kong, China
- Apollo Gleneagles Hospitals, Kolkata, India
- National University Hospital, Singapore, Singapore

REFERENCES:
- [Background] Phee SJ, Sun Z, Wang Z, Wong JY, Ho KY. The future of transluminal surgery. Expert Rev Med Devices. 2011 Nov;8(6):669-71. doi: 10.1586/erd.11.54. No abstract available. PMID 22029463
- [Background] Sun Z, Ang RY, Lim EW, Wang Z, Ho KY, Phee SJ. Enhancement of a master-slave robotic system for natural orifice transluminal endoscopic surgery. Ann Acad Med Singap. 2011 May;40(5):223-30. PMID 21678013
- [Background] Ho KY, Phee SJ, Shabbir A, Low SC, Huynh VA, Kencana AP, Yang K, Lomanto D, So BY, Wong YY, Chung SC. Endoscopic submucosal dissection of gastric lesions by using a Master and Slave Transluminal Endoscopic Robot (MASTER). Gastrointest Endosc. 2010 Sep;72(3):593-9. doi: 10.1016/j.gie.2010.04.009. Epub 2010 Jun 19. PMID 20646698
- [Background] Phee SJ, Low SC, Huynh VA, Kencana AP, Sun ZL, Yang K. Master and slave transluminal endoscopic robot (MASTER) for natural orifice transluminal endoscopic surgery (NOTES). Annu Int Conf IEEE Eng Med Biol Soc. 2009;2009:1192-5. doi: 10.1109/IEMBS.2009.5333413. PMID 19963992
- [Background] Phee SJ, Low SC, Sun ZL, Ho KY, Huang WM, Thant ZM. Robotic system for no-scar gastrointestinal surgery. Int J Med Robot. 2008 Mar;4(1):15-22. doi: 10.1002/rcs.179. PMID 18314917
- [Background] Phee SJ, Ho KY, Lomanto D, Low SC, Huynh VA, Kencana AP, Yang K, Sun ZL, Chung SC. Natural orifice transgastric endoscopic wedge hepatic resection in an experimental model using an intuitively controlled master and slave transluminal endoscopic robot (MASTER). Surg Endosc. 2010 Sep;24(9):2293-8. doi: 10.1007/s00464-010-0955-8. Epub 2010 Feb 23. PMID 20177915